CLINICAL TRIAL: NCT06098287
Title: Cost-effective Approaches to Upgrading Residential Mechanical Ventilation Systems to Control Indoor Pollutants of Both Indoor and Outdoor Origin and Improve Asthma-related Health Outcomes
Brief Title: Residential Ventilation Systems and Filtration for Asthma Control in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illinois Institute of Technology (Other)
Collaborators: Elevate (Unknown)
Responsible Party: Principal Investigator, Brent Stephens, Professor and Department Chair, Illinois Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT IRB2019-001; ILHHU0031-16 (Other Grant/Funding Number: U.S. Department of Housing and Urban Development); P-0136 (Other Grant/Funding Number: ComEd)
Record Dates: First submitted 2023-10-14; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Asthma; Pollution; Exposure
Keywords: Adult asthma; Home intervention; Mechanical ventilation; Air filtration; Indoor air pollution exposures
MeSH Terms: conditions — Asthma | interventions — Expiratory Reserve Volume

STUDY DESIGN:
Intervention Model Description: A quasi-randomized, within-subjects, parallel-group, pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Exhaust-only ventilation) (Active Comparator): A study group with a continuous exhaust-only ventilation system
  Interventions: Device: Residential mechanical ventilation system (Exhaust)
- Intervention (Central-fan-integrated-supply ventilation) (Active Comparator): A study group with an intermittent central-fan-integrated-supply ventilation system and air filtration upgrades
  Interventions: Device: Residential mechanical ventilation system (CFIS) and air filtration upgrades
- Intervention (Balanced energy recovery ventilation) (Active Comparator): A study group with a continuous balanced energy recovery ventilation system and air filtration upgrades
  Interventions: Device: Residential mechanical ventilation system (ERV) and air filtration upgrades

INTERVENTIONS:
Device: Residential mechanical ventilation system (Exhaust) — Exhaust-only ventilation system
  Arms: Intervention (Exhaust-only ventilation)
Device: Residential mechanical ventilation system (CFIS) and air filtration upgrades — Central-fan-integrated-supply ventilation system and air filtration upgrades (MERV 10)
  Arms: Intervention (Central-fan-integrated-supply ventilation)
Device: Residential mechanical ventilation system (ERV) and air filtration upgrades — Balanced energy recovery ventilation system and air filtration upgrades (MERV 10)
  Arms: Intervention (Balanced energy recovery ventilation)

SUMMARY:
The goal of this study was to investigate the effectiveness of three common approaches to upgrading residential mechanical ventilation systems in existing homes for improving asthma-related health outcomes, reducing indoor pollutants of both indoor and outdoor origin, and maintaining adequate environmental conditions and ventilation rates in a cohort of adult asthmatics in existing homes in Chicago, IL.

DETAILED DESCRIPTION:
The Breathe Easy Study utilized a quasi-randomized, within-subjects, parallel-group, pre-post intervention study design with four weeklong periods of indoor air quality (IAQ) and indoor environmental data collection for approximately one year before the installation of mechanical ventilation systems, followed by four weeklong periods of IAQ and indoor environmental data collection for approximately one year after the installation of mechanical ventilation systems, conducted from July 2017 through March 2020 in Chicago, IL. With the nature of a healthy home intervention study by installing residential mechanical ventilation systems within the timeframe, each participant received interventions in the middle of the study period, including continuous exhaust-only systems; intermittent powered central-fan-integrated-supply (CFIS) systems; or continuous balanced systems with an energy recovery ventilator. Thus, each participant served as their own control and there was no formal control group that did not receive intervention nor did they receive a sham/placebo intervention. Primary health outcome, asthma control, was assessed by using the Asthma Control Test (ACT) every month, and quality of life, stress, and other asthma-related health outcomes were assessed via the baseline and end-line surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 90+ years.
* English speaking and writing.
* Able to provide consent.
* Chicago resident.
* Households with at least one occupant with asthma
* Non-smoking houses
* Participant-owned houses
* Participant's agreement to surveys and IAQ monitoring over 2 years

Exclusion Criteria:

* Houses outside Chicago, IL USA
* Houses with significant health and safety issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Asthma Control | Each month throughout the study completion, an average of 2 years (24 months)
  Asthma Control Test (ACT) is a 5-item clinically validated survey, which is designed to measure the multi-dimensional nature of asthma control, including asthma symptoms, utilization of rescue medications, and the impact of asthma on daily functioning. The ACT score ranges from 5 ("poor control of asthma") to 25 ("complete control of asthma")

SECONDARY OUTCOMES:
Health-Related Quality of Life | Baseline (July 2017) and end-line (March 2020, end of study completion)
  12-Item Short Form Survey (SF-12) measures eight concepts commonly represented in widely used surveys: general health, physical functioning, bodily pain, vitality (energy/fatigue), social functioning, role limitations due to physical and emotional problems, and mental health (psychological distress and psychological well-being). Both the SF-12 physical (PCS) and mental (MCS) component summary scales use norm-based scoring, 0-100, with higher scores indicating better physical and mental health functioning.
Stress | Baseline (July 2017) and end-line (March 2020, end of study completion)
  Perceived Stress Scale (PSS) is a 10-item psychological assessment to understand how unpredictable, uncontrollable, and overloaded participants find their lives. The PSS score ranges from 0 to 40 with higher scores indicating higher perceived stress, and scores ranging from 0 to 13, from 14 to 26, and from 27 to 40 are considered low, moderate, and high perceived stress, respectively.
Asthma medications | Baseline (July 2017) and end-line (March 2020, end of study completion)
  Asthma medications via survey
Comorbidities | Baseline (July 2017) and end-line (March 2020, end of study completion)
  Comorbidities via survey

CONTACTS AND LOCATIONS:
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No